CLINICAL TRIAL: NCT04612894
Title: The Efficacy and Safety of Anti-PD-1 Antibody Camrelizumab Combined With Apatinib for Neoadjuvant Therapy in Locally Advanced Thyroid Cancer: a Phase II Study
Brief Title: Camrelizumab and Apatinib for Neoadjuvant Therapy in Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALA-TC
Record Dates: First submitted 2020-10-30; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; locally advanced; neoadjuvant; Camrelizumab; Apatinib
MeSH Terms: conditions — Thyroid Neoplasms | interventions — camrelizumab; apatinib; Surgical Procedures, Operative; Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Camrelizumab + Apatinib (Experimental): Apatinib 250mg, po qd, and Camrelizumab 200mg, iv q2w as neoadjuvant treatment. 28 days as one cycle, for at least two cycles.
  Interventions: Drug: Camrelizumab and Apatinib; Procedure: surgery; Procedure: core needle biopsy

INTERVENTIONS:
Drug: Camrelizumab and Apatinib — All patients will receive Camrelizumab and Apatinib for at least two cycles of neoadjuvant treatment
Procedure: surgery — Perform surgery if operable after neoadjuvant therapy
Procedure: core needle biopsy — Perform core needle biopsy if inoperable after neoadjuvant therapy

SUMMARY:
To determine the efficacy and safety of anti-PD-1 antibody Camrelizumab combined with Apatinib for neoadjuvant therapy in locally advanced thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteered to participate in the study and signed an informed consent form;
* Pathologically diagnosed locally advanced thyroid cancer, including papillary thyroid cancer, medullary cancer, follicular cancer, poorly differentiated cancer, etc., require surgical resection with or without distant metastasis;
* Preoperative assessment of locally advanced thyroid cancer (unable to achieve R0/1 resection or T4 disease);
* Have at least one measurable lesion (RECIST 1.1);
* Age>=14 years, Eastern Cooperative Oncology Group (ECOG) score 0-1;
* Patient agree to receive surgery/ core needle biopsy before and after neoadjuvant treatment.
* The main organ functions meet the criteria before treatment.

Exclusion Criteria:

* Patients who have previously been treated with immune checkpoint inhibitors (including but not limited to nivolizumab, pembrolizumab, teriplizumab, sintilizumab, etc.);
* Received external radiation therapy or iodine-131 therapy within the past 28 days; or planned systemic anti-tumor therapy during this study;
* Pathologically confirmed non-thyroid epithelial cell-derived malignant tumors (including lymphoma, metastatic cancer, sarcoma, etc.);
* With other uncontrolled / under treatment malignancies;
* Those who have multiple factors (such as inability to swallow) that affect oral medication;
* Patients with any severe and / or uncontrolled illness,
* Patients whose imaging showed that the tumor had invaded the important blood vessels or the researchers judged that the tumor was likely to invade important blood vessels during the subsequent study period and caused fatal bleeding;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of patients or affect patients to complete the research.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 24 weeks
  ORR

SECONDARY OUTCOMES:
R0/1 resection rate | at the time of surgery
  R0/1 resection rate if operable
Disease control rate | at the time point of 6 weeks
  DCR
Overall survival | up to 3 years
  OS
Adverse Events | from the first drug administration to within 90 days after surgery
  AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No